CLINICAL TRIAL: NCT05730582
Title: Increasing Uptake of EHR-enabled Population Health Outreach Strategies to Improve Diabetes Screening
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Michael Edward Bowen, Associate Professor of Internal Medicine and Pediatrics, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STU 2022-0996; R01MD016101 (NIH)
Record Dates: First submitted 2023-01-11; First posted 2023-02-16 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2; Pre Diabetes
Keywords: Diagnostic Screening Program; Health System Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Generic Screening Invitation (Active Comparator): Patients randomized to this study arm will receive the generic letter to inform them that they are at risk for T2D and that they are not up to date on screening. The letter also informs them that a screening test has been ordered, and requests that they complete testing at their clinic lab. The letter is signed by the patient's primary care provider and sent in both English and Spanish. This letter was previously developed and has been in use by the Parkland Diabetes Detection Program.
  Interventions: Behavioral: Parkland Diabetes Detection Program (PDDP) Screening Invitation
- Targeted-Tailored Screening Invitation (Experimental): Patients randomized to this study arm will receive the tailored letter, which uses messaging developed collaboratively by patients and clinical stakeholders under a prior NIH-funded research study (STU 2021-0743), in addition to available EHR data, to inform patients that they are at risk for Type 2 Diabetes based on specific clinical characteristics and that they are not up to date on screening. The letter also informs them that a screening test has been ordered, and requests that they fast and complete testing at their clinic lab within 60 days. Fasting instructions will specify nothing to eat or drink except water for at least 8 hours. The letter will be signed electronically by the patient's primary care provider and sent in both English and Spanish.
  Interventions: Behavioral: Parkland Diabetes Detection Program (PDDP) Screening Invitation
- Standard of Care (No Intervention): Patients randomized to this study arm will receive opportunistic screening based on routine clinical activities. Patients will be assigned a study number for tracking purposes, but no intervention activities via the Parkland Dysglycemia Detection Program will occur for this study arm.

INTERVENTIONS:
Behavioral: Parkland Diabetes Detection Program (PDDP) Screening Invitation — The PDDP is designed to supplement and close screening gaps that persist despite opportunistic screening. Program staff order diabetes screening tests for randomized patients, then mail screening invitation letters to inform patients that they are at risk for diabetes. The letter informs them that a screening test has been ordered, and requests that they complete testing at their clinic lab. Patients who were mailed the letter but have not completed screening after 30 days are tracked and are send a second "reminder" invitation. Patients randomized to the targeted-tailored intervention study arm receive an additional phone call after 30 days.
  Arms: Generic Screening Invitation; Targeted-Tailored Screening Invitation

SUMMARY:
The study team's central hypothesis is that the Parkland Diabetes Detection Program (PDDP) screening invitations targeted by race/ethnicity with culturally concordant messaging and tailored by glycemic risk (known PDM vs. unknown glycemic state) plus phone-based navigation of non-responders will be more effective at closing screening gaps than PDDP generic screening invitations and usual care, opportunistic screening alone.

DETAILED DESCRIPTION:
The research team will conduct a pragmatic, split cluster randomized controlled trial (clinic=cluster; patient randomization) in 12 community-based primary care clinics in an integrated safety net health system serving a high-risk, racially/ethnically diverse population.

ELIGIBILITY:
Inclusion Criteria:

* Patient is alive at time of data extraction
* Age >= 18 at time of data extraction and <76
* Visit with PCP at Parkland clinic in the last 18 months (548 days), where Encounter type = Virtual Visit or Encounter type = Office Visit
* Patient NOT included in Parkland Diabetes Registry
* Preferred language is Spanish or English
* Ethnicity is Hispanic or Non-Hispanic
* Race is White or Black
* Patient is not pregnant in last 12 months

Exclusion Criteria for Study Population 1: Prediabetes Glycemic Risk Group

* Last A1C value <5.7 (normal)
* Last A1C value >6.4 (diabetes)
* Last A1C value = blank (unchecked)
* Last A1C date occurred within last 12 months from date of export

Exclusion Criteria for Study Population 2: Score-Based Glycemic Risk Group

* Risk score <9
* Last A1C date occurred in last 30 months from date of export
* Last A1C value was >5.7 (PDM/DM)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500000 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Invitation efficacy | 60 days
  Invitation efficacy will be assessed by comparing the proportion of patients completing HgA1c or Fasting Blood Glucose screening tests at Day 60 in the targeted-tailored invitation intervention compared to the generic invitation intervention.
Program effectiveness | 12 months
  Program effectiveness will be assessed by comparing the proportion of patients completing HgA1c or Fasting Blood Glucose screening tests at Day 365 across intervention and control arms.
Direct costs | 12 months
  Direct costs of diabetes screening compared across study arms
Cost effectiveness as measured by costs per patient screened | 12 months
  Cost effectiveness will be assessed by comparing the costs per patient screened across study arms
Cost effectiveness as measured by cost per case found | 12 months
  Cost effectiveness will be assessed by comparing the costs per case found across study arms

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bowen, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No